CLINICAL TRIAL: NCT01220934
Title: Clinical Practice Surveillance of the Use of Herceptin in Patients With HER2-positive Advanced Adenocarcinoma of the Stomach or Gastro-esophageal Junction (GEJ) (HERMES)
Brief Title: An Observational Study of Herceptin (Trastuzumab) in Patients With HER2-positive Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22834
Record Dates: First submitted 2010-09-28; First posted 2010-10-14 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, multicenter study will assess the efficacy and safety of Herceptin (trastuzumab) in routine clinical practice in patients with HER2-positive advanced adenocarcinoma of the stomach or gastro-esophageal junction. Data from patients will be collected for approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Histologically confirmed advanced adenocarcinoma of the stomach or gastro-esophageal junction (GEJ) with locally advanced and/or metastatic disease
* HER2-positive tumor
* Patients who are eligible for treatment with Herceptin according to the judgment of the physician

Exclusion Criteria:

* Unwilling or unable to sign informed consent form
* Any contraindications, interactions and incompatibilities to Herceptin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastric cancer patients receiving Herceptin in routine clinical practice
Sampling Method: Probability Sample
Enrollment: 443 (Actual)
Dates: Start 2010-04-16 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Response rate according to Response Evaluation Criteria in Solid Tumors (RECIST) | 12 months
Progression-free survival according to Response Evaluation Criteria in Solid Tumors (RECIST) | 12 months
Overall survival according to Response Evaluation Criteria in Solid Tumors (RECIST) | 12 months

SECONDARY OUTCOMES:
Documentation of the testing process for HER2-positive tumors | 12 months
Assessment of implementation of guidelines and recommendations of Herceptin administration in routine clinical practice | 12 months
Documentation of backbone chemotherapy treatment and concomitant medication | 12 months
Quality of Life questionnaire | 12 months
Surveillance of pain intensity and analgesic consumption | 12 months
Surveillance of weight change | 12 months
Safety (incidence of adverse events) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Krankenhaus Nordwest; Klinik f. Onkologie und Hämatologie, Frankfurt, Germany